CLINICAL TRIAL: NCT04066582
Title: Early Feasibility Study: Application of OCT Imaging in Dermatology
Status: Completed | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: Apollo Medical Optics, Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 17CT062Be
Record Dates: First submitted 2019-08-19; First posted 2019-08-26 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Skin Diseases
Keywords: optical coherence tomography (OCT); dermatology; skin diseases; pathology; H&E stain
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Suspected skin inflammations or skin tumors
  Interventions: Device: ApolloVue™ S100 image system, Viper1-S003

INTERVENTIONS:
Device: ApolloVue™ S100 image system, Viper1-S003 — The device is an in vivo non-invasive optical coherence tomography and will be used to obtain at least 6 medical images of normal and lesional skin, respectively, for experimental group.

SUMMARY:
Optical coherence tomography (OCT) is an established medical imaging technique that uses light to capture biological images from within optical scattering media (e.g., biological tissue). A high-resolution OCT has the characteristics of non-invasive, label-free, real-time, cellular resolution with high tissue penetration depth that are highly valuable for clinical use.

AMO has developed an in-vivo OCT scanning system prototype based on the clinical needs and potential applications. This study is designed as an early feasibility study aiming for validation of AMO's in-vivo OCT scanning system in dermatology through collaboration with Mackay Memorial Hospital. The OCT can provide cellular-resolution (<1μm in lateral and axial directions) images which can be utilized to identify organelles. A high-resolution OCT has the characteristics of non-invasive, label-free, real-time, cellular resolution with high tissue penetration depth that are highly valuable for clinical use.

The proposed scenario in this study is to collecting OCT images of skins with suspicious lesion including tumor, inflammatory diseases or pigment alteration as well as normal skin by using AMO's in vivo OCT imaging system. By using traditional pathological biopsy images or dermoscopic images as gold standard references, investigators will try to identify different characteristics in OCT images of skin with suspicious lesion including tumor, inflammatory diseases, or pigment alteration as well as normal skins.

ELIGIBILITY:
Inclusion Criteria:

* A patient who is fully aware of the trial and can sign the inform consent form himself/herself
* Patients with suspected skin tumors or skin inflammations
* Patients diagnosed for biopsy
* Patients with no open wounds in the tumor or inflamed position

Exclusion Criteria:

* Patients with a transcutaneous infectious disease
* Patients under the age of 20
* Vulnerable populations, including: pregnant women, handicapped, and homelessness
* Patient cannot cooperate in examination
* Patients with skin tumors that are in the subcutaneous tissue

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population from experimental group will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects with clear tissue characteristics of skin diseases and/or normal skin in tomograms | 2 years
  Number of subjects with clear tissue characteristics of tomograms will be compared to that with unclear tissue characteristics to identify the effect of the OCT on scanning skin at study completion.
Number of subjects with the distinction between skin lesion and normal skin in tomograms | 2 years
  Number of subjects with the distinction between skin lesion and normal skin in tomograms will be compared to that with no distinction to verify the specific diseases that can be distinguished from others by the OCT at study completion.

SECONDARY OUTCOMES:
Number of subjects with clear tissue stratification of skin diseases and/or normal skin in tomograms | 2 years
  Number of subjects with clear tissue stratification, eg. dermal-epidermal junction, of tomograms will be compared to that with unclear tissue stratification to identify the effect of the OCT on scanning skin at study completion.
Number of subjects with the similarity of tissue characteristics, tissue stratification, and tissue thickness between tomograms and H&E stain | 2 years
  Number of subjects with the similarity of tissue characteristics, tissue stratification, and tissue thickness between tomograms and H&E stain will be compared to that with no similarity to verify whether the tomograms are comparable with gold standard methods H&E stain images at study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Jen Wang, MD, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, New Taipei City, Tamsui District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chang CK, Tsai CC, Hsu WY, Chen JS, Liao YH, Sheen YS, Hong JB, Lin MY, Tjiu JW, Huang SL. Errata: Segmentation of nucleus and cytoplasm of a single cell in three-dimensional tomogram using optical coherence tomography. J Biomed Opt. 2017 Mar 1;22(3):39801. doi: 10.1117/1.JBO.22.3.039801. No abstract available. PMID 28300273
- [Background] Chiu YK, Chen WL, Tsai CT, Yang CH, and Huang SL. A high en-face resolution AS-OCT providing quantitative ability to measure layered corneal opacities. European Conferences on Biomedical Optics, Munich Germany, 25-29, 2017.
- [Background] Wang SC, Hsu CY, Yang TT, Jheng DY, Yang TI, Ho TS, Huang SL. Laser-diode pumped glass-clad Ti:sapphire crystal fiber laser. Opt Lett. 2016 Jul 15;41(14):3217-20. doi: 10.1364/OL.41.003217. PMID 27420499
- [Background] Wang SC, Yang TI, Jheng DY, Hsu CY, Yang TT, Ho TS, Huang SL. Broadband and high-brightness light source: glass-clad Ti:sapphire crystal fiber. Opt Lett. 2015 Dec 1;40(23):5594-7. doi: 10.1364/OL.40.005594. PMID 26625059
- [Background] Tsai CC, Chang CK, Hsu KY, Ho TS, Lin MY, Tjiu JW, Huang SL. Full-depth epidermis tomography using a Mirau-based full-field optical coherence tomography. Biomed Opt Express. 2014 Aug 8;5(9):3001-10. doi: 10.1364/BOE.5.003001. eCollection 2014 Sep 1. PMID 25401013
- [Background] Ho TS, Yeh P, Tsai CC, Hsu KY, Huang SL. Spectroscopic measurement of absorptive thin films by spectral-domain optical coherence tomography. Opt Express. 2014 Mar 10;22(5):5675-83. doi: 10.1364/OE.22.005675. PMID 24663908
- [Background] Cheng NC, Hsieh TH, Wang YT, Lai CC, Chang CK, Lin MY, Huang DW, Tjiu JW, Huang SL. Cell death detection by quantitative three-dimensional single-cell tomography. Biomed Opt Express. 2012 Sep 1;3(9):2111-20. doi: 10.1364/BOE.3.002111. Epub 2012 Aug 13. PMID 23024905
- [Result] Wang YJ, Huang YK, Wang JY, Wu YH. In vivo characterization of large cell acanthoma by cellular resolution optical coherent tomography. Photodiagnosis Photodyn Ther. 2019 Jun;26:199-202. doi: 10.1016/j.pdpdt.2019.03.020. Epub 2019 Mar 30. No abstract available. PMID 30940575